CLINICAL TRIAL: NCT06087107
Title: Comparative Effects Of High Intensity Spinal Decompression Exercises And Eldoa On Pain, Range Of Motion And Disability In Patients Of Lumbar Radiculopathy
Brief Title: Comparative Effects Of High Intensity Spinal Decompression Exercises And Eldoa In Patients Of Lumbar Radiculopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0160 Usman Ejaz
Record Dates: First submitted 2023-10-11; First posted 2023-10-17 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Lumbar Radiculopathy
Keywords: Radiculopathy; Decompression; Pain; Range of motion
MeSH Terms: conditions — Radiculopathy; Pain

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of the treatment arms at the beginning of the trial and continue in that arm throughout the length of the trial.
Who Masked: Outcomes Assessor
Masking Description: single blinding
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Intensity Spinal Decompression Exercises (Experimental): Participants in this group will receive high intensity spinal decompression exercises
  Interventions: Other: High Intensity Spinal Decompression Exercises
- Eldoa (Active Comparator): Participants in this group will receive Eldoa.
  Interventions: Other: Eldoa

INTERVENTIONS:
Other: High Intensity Spinal Decompression Exercises — The duration of the intervention will be 4 weeks, 3 sessions a week, a total of 12 sessions will be given to the study participants. Each session will last for 40 minutes with 8-10 repetitions of each exercise.
  Arms: High Intensity Spinal Decompression Exercises
Other: Eldoa — The duration of the intervention will be 4 weeks, 3 sessions a week, and a total of 12 sessions will be given to the study participants. Each session will last for 40 minutes.
  Arms: Eldoa

SUMMARY:
To compare the effects of high intensity spinal decompression exercises and Eldoa on pain, ROM and Disability in patients of lumbar radiculopathy.

DETAILED DESCRIPTION:
In year 2020, a study conducted on the effect of eldoa alone and eldoa with core muscle strengthening to treat pain in patients with PIVD to determine the best treatment protocol between core muscle strengthening with and without eldoa to treat pain the numeric pain rating scale was used to measure pain. The study was done on 30 females randomly placed in two groups. The patients were treated for 3 days in a week on alternate days, for six consecutive weeks The eldoa technique was used segmentally on spine with different position as for l5-s1, patient flattens spine, curls back the toes curled back, inverses the ankles, internally rotates the hip, swings the arms up over the head while maintaining tension in same position as for l4-l5. Both reported decrease in pain intensity on NPRS at 6th week. So, results suggest that there was no significant difference between the effectiveness of techniques on reducing intensity of pain on NPRS.

In year 2021, a study conducted on effects of decompression and eldoa on pain and disability in lumbar disc protrusion. This study was done on 122 patients with the history of prolong sitting divided in two groups, one group was given decompression therapy and other group was treated with Eldoa which concluded that the pain could be significantly decreased while applying ELDOA for the patients with disc pathologies in musicians when assess pre and posttreatment. Likewise in this study, the quality of life of participants was significantly improved after the administration of ELDOA therapy.

In year 2022, RCT conducted on the effects of McKenzie extension exercise and ELDOA stretch in non-specific low back pain patients at railway general hospital, Rawalpindi and IRADA rehabilitation center. 48 female participants with the age range of 40-69 years and had chronic non-specific low back pain for more than 3 months were included in the study. Both groups were assessed at baseline score of ODI, BMI, NPRs after 2nd week and 4th week. According to this , McKenzie extension exercises significantly improved nonspecific low back pain and lumbar extension ROM.

In year 2022, a study conducted on effects of ELDOA Technique with Conservative Treatment on Pain Threshold of Active Trigger Points in Upper Trapezius and Levator Scpulae. She included 26 participants in her study and divided it into two groups. She measured pain, range of motion and disability after treatment. After analysis, results of her study showed that eldoa approach reduced discomfort, cervical ranges and neck impairment brought on by trigger points.

There is limited literature available regarding the effects of High intensity spinal decompression exercises and ELDOA therapy in patients with lumbar radiculopathy. Previous literature did not include the side bending and rotation component of range of motion and comparison between those two techniques. Therefore, in this study effects of ELDOA therapy will be compared with spinal decompression exercise to improve pain and range of motion and function in patients with lumbar radiculopathy and also include home plan after the session.

ELIGIBILITY:
Inclusion Criteria:

* Participants pre-diagnosed with lumber radiculopathy
* Women and men between the age of 25 to 45 years
* Participants with chronic low back pain radiated to one or both legs

Exclusion Criteria:

* Diagnosed with Spinal tumour
* Diagnosed with Lumbar spine surgery
* Diagnosed with Lumbar spondylolisthesis
* Diagnosed with Fracture of lumbar spine
* Diagnosed with Ankylosing spondylitis
* Diagnosed with Pacemaker & Taking blood thinner medication

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2023-10-20 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-01-25 (Actual)

PRIMARY OUTCOMES:
Pain(NPRS) | 4th week
  Changes from the baseline 11-point NPRS is used to capture the patient's level of pain. The scale is anchored on the left with the phrase ''no pain'' and on the right with the phrase ''worst imaginable pain.'' Patients rate their current level of pain and their worst and least amount of pain in the last 24 hours. The average of the 3 ratings or any single rating may be used to represent the patient's level of pain. Numeric pain scales have been shown to be valid and reliable with validity range from 0.86 to 0.95 and reliability r=0.96 and 0.95 with intraclass correlation coefficient of 0.95
Range of motion spine (flexion) | 4th week
  Changes from baseline ROM range of motion of spinal flexion will be taken with the help of inclinometer
Range of Motion Spine (Extension) | 4th week
  Changes from baseline ROM range of motion of spinal extension will be taken with the help of inclinometer
Range of Motion Spine (Right side bending) | 4th week
  Changes from baseline ROM range of motion of spinal right side bending will be taken with the help of inclinometer
Range of Motion Spine (left side bending) | 4th week
  Changes from baseline ROM range of motion of spinal left side bending will be taken with the help of inclinometer
Range of Motion Spine (right side rotation) | 4th week
  Changes from baseline ROM range of motion of spinal right side rotation will be taken with the help of inclinometer
Range of Motion Spine (left side rotation) | 4th week
  Changes from baseline ROM range of motion of spinal left side rotation will be taken with the help of inclinometer
Disability: Oswestry disability index questionnaire (ODI) | 4th week
  Changes from baseline ODI.is an extremely important tool that researchers and disability evaluators use to measure a patient's permanent functional disability. The test is considered the 'gold standard' of low back functional outcome tools interpretation of score are mentioned in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Faiza Amjad, MPhil, Principal Investigator — Riphah International University
Locations (1):
- Ittefaq hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Iversen T, Solberg TK, Wilsgaard T, Waterloo K, Brox JI, Ingebrigtsen T. Outcome prediction in chronic unilateral lumbar radiculopathy: prospective cohort study. BMC Musculoskelet Disord. 2015 Feb 7;16(1):17. doi: 10.1186/s12891-015-0474-9. PMID 25887469
- [Background] Ostelo RW. Physiotherapy management of sciatica. J Physiother. 2020 Apr;66(2):83-88. doi: 10.1016/j.jphys.2020.03.005. Epub 2020 Apr 11. No abstract available. PMID 32291226
- [Background] Berry JA, Elia C, Saini HS, Miulli DE. A Review of Lumbar Radiculopathy, Diagnosis, and Treatment. Cureus. 2019 Oct 17;11(10):e5934. doi: 10.7759/cureus.5934. PMID 31788391
- [Background] Grimm BD, Blessinger BJ, Darden BV, Brigham CD, Kneisl JS, Laxer EB. Mimickers of lumbar radiculopathy. J Am Acad Orthop Surg. 2015 Jan;23(1):7-17. doi: 10.5435/JAAOS-23-01-7. PMID 25538126